CLINICAL TRIAL: NCT05074524
Title: Evaluating Repetitive Transcranial Magnetic Stimulation to Reduce Opioid Cravings in Adults Who Use Heroin
Brief Title: Repetitive Transcranial Magnetic Stimulation to Reduce Heroin Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Hyunhwa Lee, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1748113-2
Record Dates: First submitted 2021-07-30; First posted 2021-10-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Opioid-use Disorder; Heroin Abuse; Craving; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rTMS group (Experimental): Active rTMS treatment will be delivered at 10 Hz, 100% resting motor threshold, 2000 pulses delivered in five seconds per train with 10-second intra-train pause, delivered once daily five days per week, Monday through Friday for 10 days (10 total treatments). This protocol is adapted from Shen and colleagues (2016), who did not report any adverse events. Liu and colleagues (2020) also used the same protocol and only reported mild side effects of dizziness, headache, and insomnia, which resolved by the 30-day follow-up. However, it is unclear whether these side effects resolved sooner than the 30-day follow-up.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Placebo Group (Sham Comparator): The control group will undergo the same seat positioning and comfort measures but will not have a resting motor threshold determination. The coil will be turned 90 degrees counter-clockwise, and the side of the coil will rest on the scalp over the area of the skull corresponding to the motor cortex, so the participant will feel the coil making contact. The same treatment protocol in the active rTMS group will be initiated to mimic the sound of rTMS treatment, though no pulses will be delivered to the participant because of the coil rotation.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Active rTMS treatment will be delivered at 10 Hz, 100% resting motor threshold, 2000 pulses delivered in five seconds per train with 10-second intra-train pause, delivered once daily five days per week, Monday through Friday for 10 days (10 total treatments). This protocol is adapted from Shen and colleagues (2016), who did not report any adverse events. Liu and colleagues (2020) also used the same protocol and only reported mild side effects of dizziness, headache, and insomnia, which resolved by the 30-day follow-up. However, it is unclear whether these side effects resolved sooner than the 30-day follow-up.
  Arms: rTMS group
Device: Sham Repetitive Transcranial Magnetic Stimulation — The control group will undergo the same seat positioning and comfort measures but will not have a resting motor threshold determination. The coil will be turned 90 degrees counter-clockwise, and the side of the coil will rest on the scalp over the area of the skull corresponding to the motor cortex, so the participant will feel the coil making contact. The same treatment protocol in the active rTMS group will be initiated to mimic the sound of rTMS treatment, though no pulses will be delivered to the participant because of the coil rotation.
  Arms: Placebo Group

SUMMARY:
The purpose of this research study is to test the effect of repetitive transcranial magnetic stimulation (rTMS) on opioid cravings among adult patients with Opioid Use Disorder.

DETAILED DESCRIPTION:
This study will use rTMS, a neuromagnetic and non-invasive treatment, to reduce opioid cravings in individuals who are diagnosed with opioid use disorder. Repetitive transcranial magnetic stimulation is currently used for the treatment of Major Depressive Disorder and Obsessive Compulsive Disorder in clinical practice. This proposed study will employ a randomized, single-blind, experimental design. Participants will be randomly assigned to two groups using a computer-based randomization program: treatment and sham-control groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-64, used heroin in the past 30 days;
* has a history of heroin use for at least one year;
* meets the clinical criteria for Opioid Use Disorder (only heroin use will be considered to meet this criteria);
* meets the clinician clearance using the rTMS Patient Screening Form.

Exclusion Criteria:

* do not currently take and medications for a substance use disorder such as methadone, buprenorphine, naltrexone, acamprosate, disulfiram;
* do not have a psychotic disorder;
* do not have a diagnosis of another substance use disorder;
* do not have a history of seizures or other neurological disorders including organic brain disease; epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery;
* do not have a personal history of head trauma that resulted in a loss of consciousness for more than 5 minutes and retrograde amnesia for more than 30 minutes;
* do not have a presence of non-fixed metal in body 30 cm to treatment coil.
* have not taken any medication for a substance use disorder within the last 72 hours before the first rTMS treatment;
* are not pregnant or think you may be pregnant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Desires for Drug Questionnaire | Days 1, 3, 5, 8, 10, 12, 42
  This standardized questionnaire measures cravings for opioids. This scale includes a total of 13 items. Scoring is based on a 1-7 likert scale for each item. Specific items are assigned to one of three domains: desire, negative reinforcement, and control. A higher score indicates higher level of cravings. A lower score indicates a lesser level of opioid cravings, which is a better outcome. The primary outcome measure will be measured at various time points throughout the study to assess a change.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No